CLINICAL TRIAL: NCT05556473
Title: A Pilot Study of 1-(2-[18f]Fluoroethyl)-L-Tryptophan PET/CT Imaging In Human Cancers
Brief Title: F-Tryptophan PET/CT in Human Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Csaba Juhasz, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-010
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Glioma; Metastatic Brain Tumor; Breast Cancer; Neuroendocrine Tumors; Rectal Cancer
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Neuroendocrine Tumors; Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]FETrp PET radiotracer (Experimental): All participants will receive the tracer to evaluate the uptake of [18F]FETrp PET/CT on intra- and extracranial cancers.
  Interventions: Drug: 1-(2-[18F]FLUOROETHYL)-L-Tryptophan

INTERVENTIONS:
Drug: 1-(2-[18F]FLUOROETHYL)-L-Tryptophan — Radioactive tracer 1-(2-[18F]FLUOROETHYL)-L-Tryptophan 0.14mCi/kg/5MBq/kg injection given one time prior to PET Scan.
  Other Names: [18F]FETrp PET radiotracer

SUMMARY:
Imaging procedures such as 1-(2-[18F]FLUOROETHYL)-L-Tryptophan PET/CT in patients with cancers may help doctors assess a patient's response to treatment and help plan the best treatment in the future. The purpose is to see if there can be a better differentiation of tumor and non-tumor tissue where the tumor tissue has a higher uptake of Tryptophan.

DETAILED DESCRIPTION:
In this research study, we will compare the uptake of the tracer on F-Tryp PET/CT in patients with cancers; specifically, to evaluate whether the tumors show increased tracer uptake as compared to non-tumor tissues, using F-Tryp PET/CT. Additionally, we will evaluate the biodistribution (i.e. track where the tracer has traveled in the body) and radiation dosimetry (i.e., absorbed dose of tracer in tissue). These changes may be compared with results of the physical examination and scans (CT and MRI or standard clinical PET) that are done as part of routine clinical care or as part of other studies. Pictures (images) from the PET scan will be made showing the distribution throughout the body of substances containing a small amount of radioactive material.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Targeted lesion (tumor) is at least 1 cm in diameter as shown by clinical imaging.
* Patient is able to lie in the PET/CT scanner for at least 70 minutes while undergoing scanning.
* Women of childbearing potential must not be pregnant or breastfeeding.
* Recent anatomic imaging with visible disease (tumor) for comparison with the PET/CT. .
* Physical exam within 28 days of PET imaging, CBC and Multiphasic (including electrolytes, BUN, creatinine, total bilirubin, AST and ALT) within 14 days.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

Inclusion Criteria Specific for Intracranial Tumors

- Clinical and MRI diagnosis of an intracranial lesion suspicious for a brain tumor, including gliomas or metastatic brain tumors; primary, residual, or recurrent brain tumors (judged by clinical imaging) will qualify.

Inclusion Criteria Specific for Extracranial Neuroendocrine Tumors:

* Histopathologically confirmed, well-differentiated metastatic neuroendocrine tumor.
* ECOG performance status of 2 or better.
* Patients receiving stable-dose somatostatin analogs (SSAs, long-acting release [LAR], depot) for >3 months before enrollment may be enrolled on the study, but such treatment is not required.

Inclusion Criteria specific for Extracranial Primary Breast tumors:

* Clinical and radiological diagnosis of a breast cancer
* ECOG performance status of 2 or better.

Inclusion Criteria specific for Rectal tumors:

* Histologically confirmed colorectal cancer, which is located in the rectum.
* ECOG performance status of 2 or better.

Exclusion Criteria:

* Patients who are pregnant or lactating are excluded.

Exclusion Criteria Specific for Intracranial Tumors:

* Severe increased intracranial pressure, status epilepticus, or other symptoms requiring emergency or urgent intervention.
* Tumor surgery or radiation within 1 month prior to the PET scan

Exclusion Criteria Specific for Extracranial Neuroendocrine Tumors:

* Tumor-directed therapy within 3 months to the area of planned imaging.
* Ongoing treatment with a targeted agent (e.g., sunitinib or everolimus) or receiving cytotoxic chemotherapy (e.g., capecitabine or temozolomide).
* Use of telotristat ethyl (a tryptophan-hydroxylase inhibitor) within one month.

Exclusion Criteria for Extracranial Primary Breast tumors:

-Recent (within 1 month) tumor resection or radio-chemotherapy (acute/subacute post-treatment inflammatory changes may cause false positive increases on PET).

Exclusion Criteria for Rectal tumors:

-Active inflammatory bowel disease (Crohn's or Ulcerative colitis) involving the rectum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The percent difference in tracer uptake values between the tumor mass and the background (non-tumor tissue) | During procedure (from right after tracer injection to 1-hour post-injection)
  The percent difference in 1-(2-[18F]fluoroethyl)-L-tryptophan tracer standardized uptake values, measured between tumor and non-tumor (normal) tissues by PET/CT imaging, in each subject, will be calculated. Mean and standard deviation of the percent differences will be calculated for each tumor type.
Correlation between the 1-(2-[18F]fluoroethyl)-L-tryptophan tracer uptake values and the tracer transport rates measured in the same breast tumor tissue. | During procedure (from right after tracer injection to 1-hour post-injection)
  The 1-(2-[18F]fluoroethyl)-L-tryptophan tracer standardized uptake values and the volume of distribution (characterizing the tracer transport rates) will be measured by PET/CT imaging in the same breast tumor tissues, and the correlation of these two measures will be calculated.

SECONDARY OUTCOMES:
Radiation doses to the various organs. | During procedure (from right after tracer injection to 1-hour post-injection)
  Radiation doses received by the various organs (heart, lungs, pancreas, gallbladder, liver, small intestines, kidneys, muscle, bladder, ovaries/testes) will be measured from the dynamic 1-(2-[18F]fluoroethyl)-L-tryptophan PET/CT images. Mean and standard deviation of the radiation doses will be calculated for each organ.
Overall radiation dose to the study participants. | During procedure (from right after tracer injection to 1-hour post-injection)
  Overall radiation dose received by the study participants from the PET/CT scan will be calculated from the dynamic 1-(2-[18F]fluoroethyl)-L-tryptophan PET/CT images. Mean and standard deviation of the overall radiation dose will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Juhasz, M.D.,Ph.D, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No